CLINICAL TRIAL: NCT05296577
Title: A Controlled, Phase II Study of Anlotinib vs Placebo Combination With Vinorelbine for the Treatment of HER2- Advanced Breast Cancer
Brief Title: Anlotinib Combination With Vinorelbine in the HER2- Advanced Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, Min Yan, MD, Chief physician, Henan Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANLO-BC
Record Dates: First submitted 2022-03-16; First posted 2022-03-25 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Breast Cancer
Keywords: anlotinib; vinorelbine; HER2 negtive; advanced
MeSH Terms: conditions — Breast Neoplasms | interventions — anlotinib; Vinorelbine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- anlotinib and vinorelbine (Experimental): anlotinib combined with vinorelbine
  Interventions: Drug: anlotinib and vinorelbine
- vinorelbine (Placebo Comparator): placebo and vinorelbine
  Interventions: Drug: Vinorelbine injection

INTERVENTIONS:
Drug: anlotinib and vinorelbine — anlotinib 12mg orally ,2 weeks on/1 week off ,Q3W; vinorelbine 25-30mg/m2 intravenously ,D1/8,21 days as a cycle.Imaging will be performed after the twice anlotinib administration as 2 cycles.
  Other Names: AL3818 and vinorelbine
  Arms: anlotinib and vinorelbine
Drug: Vinorelbine injection — vinorelbine 25-30mg/m2 intravenously ,D1/8,21 days as a cycle.Imaging will be performed after the twice anlotinib administration as 2 cycles.
  Other Names: vinorelbine
  Arms: vinorelbine

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of anlotinib combined with vinorelbine in the treatment of HER2- advanced breast cancer.

DETAILED DESCRIPTION:
The eligible patients were HER2 negative advanced breast cancer patients who experienced failure of previous treatments with anthracyclines and/or taxanes , or hormone receptor-positive HER2-negative advanced breast cancer patients who progressed after at least first-line endocrine therapy in the advanced stage.The enrolled patients would receive anlotinib 12mg orally (2 weeks on/1 week off ,Q3W) plus vinorelbine 25-30mg/m2 intravenously (D1/8,21 days as a cycle) or vinorelbine 25-30mg/m2 intravenously (D1/8,21 days as a cycle).Imaging will be performed after the twice anlotinib administration as 2 cycles.This study is a randomized controlled, phase II clinical trial, and the treatment continued until radiographic progression,unacceptable toxicity, investigator or patient decision to withdraw, non-adherence to treatment or trial procedures.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients voluntarily participated in the study and signed informed consent;
* 2. Women aged 18 or older;
* 3. The number of treatment lines shall not exceed 4 lines;
* 4. Patients with locally advanced or metastatic breast cancer diagnosed as HER2-negative by molecular typing;
* 5. Enrolled patients were HER2-negative breast cancer patients who had failed to prior taxane and/or anthracycline therapy, or patients with hormone receptor-positive HER2-negative advanced breast cancer who had progressed with at least prior first-line endocrine therapy;
* 6. ECOG score is 0 or 1, and the expected survival is not less than 3 months;
* 7. Patients with measurable lesions as defined in RECIST1.1 criteria;
* 8. The main organs function well, and the laboratory test indexes meet the following requirements:(1) Routine blood test (no blood transfusion or hematopoietic stimulating factor was used within 7 days before screening) :① Hemoglobin (HB) ≥ 90g/L;② Absolute neutrophil count (ANC) ≥1.5×109/L;③ Platelet (PLT) ≥ 80×109/L;(2) Blood biochemical test (no blood transfusion or albumin within 7 days before screening) :① ALT and AST ≤2.5 × ULN (liver/bone metastasis ≤5 × ULN; Bone metastases ≤5 ULN);② Serum total bilirubin (TBIL) ≤1.5 × ULN;③ Serum Cr≤1.5×ULN or creatinine clearance ≥60 mL /min;(3) Coagulation function test:① Activated partial thrombin time (APTT), international standardized ratio (INR), prothrombin time (PT) ≤ 1.5×ULN;② Doppler ultrasound assessment: left entricular ejection fraction (LVE F)≥ 50%;
* 9. The patient has the ability to take medication orally;
* 10. Any toxic side effects of previous chemotherapy have been recovered to ≤CTCAE1 or baseline level;
* 11. Women of reproductive age must agree to use a highly effective method of contraception during the study period and for 6 months after the last administration of the study drug; Negative serum or urine pregnancy test within 7 days prior to study enrollment and must be non-lactating subjects;

Exclusion Criteria:

* 1. Prior treatment with bevacizumab, anlotinib and other antiangiogenic agents;
* 2. Patients who had previously used Vinorelbine with an interval time of less than 6 months from the end of medication;
* 3. Interval of less than 3 weeks after radiotherapy or chemotherapy; The interval after endocrine therapy was less than 1 week;
* 4. Associated diseases/history;(1) Clinically significant hemoptysis occurred within 3 months before enrollment (hemoptysis > 50ml per day); Or bleeding symptoms of significant clinical significance or a clear bleeding tendency, such as gastrointestinal bleeding, hemorrhagic gastric ulcer, baseline fecal occultation and above, or suffering from vasculitis, etc.;(2) Arteriovenous thrombosis events occurred within 6 months before enrollment, such as cerebrovascular accident (including temporary ischemic attack), deep venous thrombosis (except those who had been cured after intravenous catheterization due to chemotherapy) and pulmonary embolism, etc.;(3) hypertension, which cannot be well controlled by antihypertensive drug therapy (systolic blood pressure & GT; 140 mmHg or diastolic pressure > 90 mmHg); During the first 6 months of randomization, myocardial infarction, severe/unstable angina, NYHA grade 2 or higher cardiac dysfunction, clinically significant ventricular arrhythmias or ventricular arrhythmias, and symptomatic congestive heart failure;(4) Interstitial lung disease, non-infectious pneumonia or uncontrollable systemic diseases (e.g., diabetes, pulmonary fibrosis and acute pneumonia);(5) Renal insufficiency: urine protein ≥ ++ indicated by routine urine examination, or confirmed 24-hour urine protein level ≥1.0g;(6) History of live attenuated vaccine vaccination within 28 days prior to initial study administration or expected live attenuated vaccine vaccination during study period;(7) human immunodeficiency virus (HIV) infection or known acquired immunodeficiency syndrome (AIDS); Active hepatitis (hepatitis B, defined as HBV-DNA ≥ 500 IU/ mL; Hepatitis C, defined as hcV-RNA higher than the lower limit of assay) or co-infection with hepatitis B and c;(8) Severe infection, including but not limited to bacteremia and severe pneumonia requiring hospitalization, occurred within 4 weeks before the first administration; Active CTCAE grade 5.0≥2 infection requiring systemic antibiotic treatment within 2 weeks prior to initial administration or unexplained fever during screening/prior to initial administration > 38.5°C (according to the investigator's judgment, fever caused by tumor can be included in the group); Evidence of active tuberculosis infection within 1 year before administration;
* 5. Have been diagnosed with any other malignant tumor within 3 years prior to entering the study;
* 6. Thyroid dysfunction;
* 7. Major operations were performed within 28 days before enrollment, and minor operations were performed within 14 days before enrollment;
* 8. Subjects who have received or are planning to receive allogeneic bone marrow transplantation or solid organ transplantation;
* 9. Peripheral neuropathy ≥ grade 2; Patients with active brain metastases, cancerous meningitis, spinal cord compression, or diseases of the brain or pia meningiae found by imaging CT or MRI examination at the time of screening (patients with brain metastases who had completed treatment 14 days before enrollment and had stable symptoms could be enrolled, but were confirmed to have no symptoms of cerebral hemorrhage by craniocerebral MRI, CT or venography evaluation);
* 10. There are significant factors affecting oral drug absorption, such as inability to swallow, chronic diarrhea, and the presence of clinically significant intestinal obstruction.
* 11. Female subjects who are pregnant, breast-feeding, or planning to become pregnant during the study period.
* 12. Patients with other serious physical or mental disorders or abnormal laboratory tests that may increase the risk of study participation or interfere with study results, and who are considered unsuitable for study participation by the investigator.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2022-03-22 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
PFS | up to 24 months
  progression-free survival

SECONDARY OUTCOMES:
ORR | up to 24 months
  Objective Response Rate
OS | up to 24 months
  overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Min Yan, Principal Investigator — Henan Cancer Hospital
Locations (1):
- Henan Cancer Hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after de-identificationare available following article publication.
Supporting Information: Study Protocol
Time Frame: five years after publication
Access Criteria: Please contact Central contact person by Email